CLINICAL TRIAL: NCT07311993
Title: A Phase 1b, Open-Label Parallel Study Evaluating CLR 125 in Patients With Relapsed or Refractory Triple Negative Breast Cancer
Brief Title: Phase 1 Study of CLR 125 in Triple Negative Breast Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Cellectar Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DCL-25-003
Record Dates: First submitted 2025-11-13; First posted 2025-12-31 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-12

CONDITIONS: Breast Cancer
Keywords: triple negative breast cancer
MeSH Terms: conditions — Breast Neoplasms; Triple Negative Breast Neoplasms | interventions — CLR1404

STUDY DESIGN:
Intervention Model Description: CLR 125 is a radio-iodinated therapy comprising a core phospholipid ether (PLE) analogue radiolabeled with iodine-125. CLR 125 exploits the tumor-targeting properties of PLEs to provide targeted delivery of Auger-emitting radiation to malignant tumor cells and minimizes radiation exposure to normal tissues.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Dosimetry Phase (Other): Iopofosine I 131 (CLR 131) will be administered at 10 mCi on day 1 for approximately 15 patients for imaging purposes.
  Interventions: Drug: Iopofosine I 131
- Treatment Phase: CLR 125 Arm 1 (Experimental): CLR 125 administered at 65 mCi/m2 fractionated over four doses (day 1, 2, 8, and 9) in each 8-week cycle; patient will receive up to 4 cycles.
  Interventions: Drug: CLR 125
- Treatment Phase: CLR 125 Arm 2 (Experimental): CLR 125 will be administered at 125 mCi/m2 fractionated over four doses (day 1, 2, 8, and 9) in each 8-week cycle; patient will receive up to 3 cycles.
  Interventions: Drug: CLR 125
- Treatment Phase: CLR 125 Arm 3 (Experimental): CLR 125 will be administered at 190 mCi/m2 fractionated over four doses (day 1, 2, 8, and 9) in each 8-week cycle; patient will receive up to 2 cycles.
  Interventions: Drug: CLR 125

INTERVENTIONS:
Drug: Iopofosine I 131 — Investigational radiopharmaceutical product intended for IV administration.
  Other Names: CLR 131
  Arms: Dosimetry Phase
Drug: CLR 125 — Investigational radiopharmaceutical product intended for IV administration.
  Arms: Treatment Phase: CLR 125 Arm 1; Treatment Phase: CLR 125 Arm 2; Treatment Phase: CLR 125 Arm 3

SUMMARY:
The goal of this clinical trial is to evaluate the safety and efficacy of 3 different dose levels of CLR 125 in patients with advanced triple negative breast cancer. The main questions the study aims to answer are:

* What dose and regimen should be used in future trials of CLR 125 in patients with advanced triple negative breast cancer.
* What side effects do participants have when taking CLR 125.

Participants will:

* Have CLR 125 administered via infusion 4 times each cycle; repeated every 8 weeks.
* Visit the clinic once every 3 weeks for checkups and testing.
* Report any side effects or new medications.

Some participants may also receive one dose of CLR 131 to evaluate the amount of radiation delivered to various organs and to the tumor. These participants will:

* Have 4 scans completed over 2 weeks
* Have blood drawn 6 times over 2 weeks.

DETAILED DESCRIPTION:
This study is designed to determine the recommended dose and regimen for future trials and to evaluate the safety and tolerability of CLR 125 at the selected doses in patients with advanced triple negative breast cancer. It will also determine the antitumor activity (treatment response by RECIST v1.1) through assessment of overall response rate, progression free survival, overall survival, duration of response and duration of clinical benefit of CLR 125 in patients with advanced triple negative breast cancer.

Total body, organ, and tumor dosimetry will be assessed in a select number of patients prior to CLR 125 dosing. At the conclusion of the study, total body, organ, and tumor dosimetry will be calculated for the intended patient population, to inform future studies.

Up to 60 evaluable patients will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Unequivocal TNBC histology [ER and PR less than 10% each and HER-2 negative].
* Patients that have progressed after at least one prior standard therapeutic regimen given alone or in combination (including, but not limited, to: chemotherapy, immunotherapy, sacituzumab govitecan-hziy, trastuzumab deruxtecan).

  * Patients who have received neo-adjuvant or adjuvant therapy must be at least one year from that treatment regimen.
* Patient is ≥ 18 years of age.
* ECOG performance status of 0 to 2.
* Life expectancy ≥ 6 months.
* Patient must meet the following laboratory criteria:

  * Platelets ≥ 75,000/uL [75 x 10^9/L]
  * White blood cell (WBC) count ≥ 3000/uL
  * Absolute neutrophil count ≥ 1500/uL
  * Hemoglobin ≥ 9 g/dL
  * Estimated glomerular filtration rate ≥ 30 mL/min/1.73 m2 (as reported by the local lab)
  * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 × upper limit of normal (ULN)
  * Bilirubin < 1.5 × ULN
* At least one measurable lesion, as defined by RECIST v1.1, with longest diameter at baseline ≥ 10 mm (excluding lymph nodes, for which the short diameter must be ≥ 15 mm).
* Patients with known brain metastases must have completed any radiotherapy or systemic treatments for brain metastases prior to enrollment; by investigator assessment be considered stable with no new signs or symptoms for at least 1 month, and on a stable dose of steroids (unchanged for three weeks prior to registration or on a steroid tapering regimen).
* Patients must express willingness and ability to comply with scheduled study visits, treatment plans, laboratory tests, and other study procedures.
* Patient or their legally authorized representative must have the ability to understand and provide signed informed written consent before the initiation of any study-related procedures.
* Female patients of childbearing potential must have a negative pregnancy test within 24 hours of dosing.
* Women of childbearing potential must agree to use a highly effective method of contraception during the study and for 12 months following administration of the study drug. Highly effective methods of contraception include combined (estrogen and progestogen containing) hormonal contraceptives associated with inhibition of ovulation, progestogen-only hormonal contraception associated with inhibition of ovulation, intrauterine device, intrauterine hormone-releasing system, vasectomized partner, or sexual abstinence. Women who have undergone hysterectomy, bilateral oophorectomy, or bilateral tubal ligation, or are post-menopausal (no menses for 12 months without an alternative medical cause) are considered to be of non-childbearing potential.
* Men who are able to father a child must agree to use a condom during the study and for 12 months following administration of the study drug.

Exclusion Criteria:

* Antitumor systemic therapy or investigational therapy, within three-half-lives of the agent preceding study drug administration. NOTE: Patients participating in non-interventional clinical trials (i.e., non-drug) are allowed to participate in this trial.

  * Focal radiation (including palliative radiation) to non-target lesions should be completed at least 2 weeks prior to dosing.
  * For patients receiving CLR 125 after participation in the dosimetry phase, CLR 131 washout is not required prior to dosing with CLR 125.
* Prior targeted radiotherapy.
* Prior external beam radiation therapy resulting in greater than 20% of total bone marrow receiving greater than 20 Gy. For estimation purposes, the following bone marrow percentages can be used:

  * Vertebral bodies: Cervical 0.5%, thoracic 1%, lumbar 2% per vertebral body
  * Hemipelvis (ilium, acetabulum, ischium): 13% per side
  * Sacrum: 10%
  * Skull: 12%
  * Scapula: 5% per side
  * Ribs: 4% per side
  * Femur: 3% per side
* Ongoing Grade 2 or greater toxicities due to previous therapies, excluding alopecia, that in the opinion of investigator might be exacerbated by study treatment.
* Patients with prior or concurrent malignancy other than TNBC with the following exceptions, which must be fully treated with no evidence of disease for at least 2 years: non-melanoma skin cancers only requiring topical treatment or surgical excision; melanoma in situ; treated cervical carcinoma in situ; successfully treated prostate cancer.
* Any other concomitant serious illness or organ system dysfunction (including cardiac and pulmonary dysfunction) that in the opinion of the Investigator would either compromise patient safety or interfere with the evaluation of the safety of the test drug.
* Known history of human immunodeficiency virus or uncontrolled, serious, active infection.
* Pregnancy or breast-feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-12-05 (Actual); Primary Completion 2028-02 (Estimated); Study Completion 2029-07 (Estimated)

PRIMARY OUTCOMES:
Dose Determination for CLR 125 | 57 days after initiation of last cycle (each cycle is 57 days)
  Identify the recommended Phase 2 dose and regimen of CLR 125 in advanced TNBC patients
Number of adverse events related to study treatment (CLR 125) | Assessed throughout the study through 1 year following completion of treatment.
  Adverse Events are graded per NCI CTCAE v5.0

SECONDARY OUTCOMES:
Efficacy Evaluation for Overall Response Rate | 57 days after initiation of last cycle (each cycle is 57 days)
  To determine the overall response (ORR) rate as assessed by RECIST v1.1.
Efficacy Evaluation for Progression Free Survival | Assessed throughout the study through 1 year following completion of treatment
  To determine the therapeutic activity defined as Progression Free Survival (PFS) using Kaplan Meier estimator.
Efficacy Evaluation for Overall Survival | Assessed throughout the study through 1 year following completion of treatment
  To determine the therapeutic activity defined as Overall Survival (OS) using Kaplan Meier estimator.
Evaluation for Duration of Response | Assessed throughout the study through 1 year following completion of treatment
  To determine the therapeutic activity defined as Duration of Response (DOR) using Kaplan Meier estimator.
Efficacy Evaluation for Duration of Clinical Benefit | Assessed throughout the study through 1 year following completion of treatment.
  To determine the therapeutic activity defined as Duration of Clinical Benefit (DOCB) using Kaplan Meier estimator.

OTHER OUTCOMES:
Dosimetry Evaluation for Total Body and Normal Organs | 1 hour post-infusion and concluding 11 days post-initial imaging
  To determine total body and organ radiation dosimetry, together, of iopofosine I 131 (CLR 131) in advanced TNBC patients
Tumor Dosimetry Evaluation of iopofosine I 131 (CLR 131) | 1 hour post-infusion and concluding 11 days post-initial imaging
  Determine the tumor dosimetry of iopofosine I 131 (CLR 131) in advanced TNBC patients.

CONTACTS AND LOCATIONS:
Overall Officials: Jarrod Longcor, Study Director — Cellectar Biosciences
Locations (2):
- United States (2):
  - Mayo Clinic Florida, Jacksonville, Florida
  - United Theranostics, Glen Burnie, Maryland

IPD SHARING:
Plan to Share IPD: No